CLINICAL TRIAL: NCT02558296
Title: A Double Blind Placebo Controlled Study to Evaluate the Effects of Bexagliflozin on Hemoglobin A1c in Patients With Type 2 Diabetes and Increased Risk of Cardiovascular Adverse Events
Brief Title: Bexagliflozin Efficacy and Safety Trial
Acronym: BEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-476
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bexagliflozin tablets, 20 mg (Active Comparator): Each subject will receive bexagliflozin 20 mg once daily for the duration of the study.
  Interventions: Drug: Bexagliflozin
- Placebo tablets (Placebo Comparator): Each subject will receive placebo (inactive tablet) once daily for the duration of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bexagliflozin — 20 mg, tablet
  Other Names: EGT0001442; EGT0001474
  Arms: Bexagliflozin tablets, 20 mg
Drug: Placebo — 20 mg tablet to match active comparator
  Arms: Placebo tablets

SUMMARY:
The purpose of this study is to investigate the effect of bexagliflozin in lowering hemoglobin A1c (HbA1c) levels in patients with type 2 diabetes mellitus (T2DM) and increased risk of cardiovascular adverse events.

The data from this study will be combined with the data from other bexagliflozin studies in a meta-analysis of CV safety outcomes.

DETAILED DESCRIPTION:
Approximately 130 investigative sites globally are planned to participate in this study.

An estimated 1650 subjects with inadequately controlled T2DM and an elevated risk of cardiovascular adverse events will be randomized to bexagliflozin tablets, 20 mg, or placebo in a ratio of 2:1 in addition to the background anti-diabetic medications.

The study is an event-driven trial. The treatment period will end when the last randomized subject has completed at least 52 weeks of treatment and a total of at least 134 subjects have experienced a cardiac event.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of T2DM
* Subjects who have had a stable treatment regimen for T2DM for the past 3 months
* Subjects who present with at least one of the following 3 histories:

Group 1: A history of atherosclerotic vascular disease Group 2: A history of heart failure Group 3: Age ≥ 55 years with diabetes for ≥ 10 years, uncontrolled hypertension, currently smoking, reduced kidney function, or cholesterol problems

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus or maturity-onset/diabetes of the young
* History of genitourinary tract infections
* Evidence of abnormal liver function
* History of MI, stroke or hospitalization for heart failure in the past 3 months
* Prior kidney transplant or evidence of kidney problems
* Prior or planned pace maker implantation
* Pregnant or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Lock, MD, Study Director — Theracos
Locations (157):
- United States (66):
  - Research Site 1090, Gilbert, Arizona
  - Research Site 1041, Little Rock, Arkansas
  - Research Site 1073, Azusa, California
  - Research Site 1076, Concord, California
  - Research Site 1078, Fresno, California
  - Research Site 1089, Harbor City, California
  - Research Site 1058, Lincoln, California
  - Research Site 1051, Los Angeles, California
  - Research Site 1004, Los Angeles, California
  - Research Site 1068, Montclair, California
  - Research Site 1077, Orange, California
  - Research Site 1218, Denver, Colorado
  - Research Site 1092, Golden, Colorado
  - Research Site 1216, Norwalk, Connecticut
  - Research Site 1083, Newark, Delaware
  - Research Site 1057, Boca Raton, Florida
  - Research Site 1059, Brooksville, Florida
  - Research Site 1050, Panama City, Florida
  - Research Site 1099, Port Charlotte, Florida
  - Research Site 1066, Tampa, Florida
  - Research Site 1072, Augusta, Georgia
  - Research Site 1082, Pocatello, Idaho
  - Research Site 1258, Champaign, Illinois
  - Research Site 1043, Anderson, Indiana
  - Research Site 1071, Avon, Indiana
  - Research Site 1086, Des Moines, Iowa
  - Research Site 1224, Covington, Kentucky
  - Research Site 1228, Annapolis, Maryland
  - Research Site 1221, Baltimore, Maryland
  - Research Site 1079, Hyattsville, Maryland
  - Research Site 1223, Midland, Michigan
  - Research Site 1217, Petoskey, Michigan
  - Research Site 1254, Ypsilanti, Michigan
  - Research Site 1054, St Louis, Missouri
  - Research Site 1060, St Louis, Missouri
  - Research Site 1252, Kalispell, Montana
  - Research Site 1052, Omaha, Nebraska
  - Research Site 1263, Omaha, Nebraska
  - Research Site 1080, Las Vegas, Nevada
  - Research Site 1219, Somerset, New Jersey
  - Research Site 1044, Albuquerque, New Mexico
  - Research Site 1220, Saratoga Springs, New York
  - Research Site 1264, The Bronx, New York
  - Research Site 1049, West Seneca, New York
  - Research Site 1085, Chapel Hill, North Carolina
  - Research Site 1074, Charlotte, North Carolina
  - Research Site 1056, Morehead City, North Carolina
  - Research Site 1229, Wilmington, North Carolina
  - Research Site 1064, Winston-Salem, North Carolina
  - Research Site 1075, Fargo, North Dakota
  - Research Site 1266, Lindsay, Oklahoma
  - Research Site 1055, Oklahoma City, Oklahoma
  - Research Site 1265, Oklahoma City, Oklahoma
  - Research Site 1046, Oklahoma City, Oklahoma
  - Research Site 1260, Lancaster, Pennsylvania
  - Research Site 1042, Cumberland, Rhode Island
  - Research Site 1225, Austin, Texas
  - Research Site 1259, Dallas, Texas
  - Research Site 1048, Kingwood, Texas
  - Research Site 1070, Lampasas, Texas
  - Research Site 1222, Lewisville, Texas
  - Research Site 1081, North Richland Hills, Texas
  - Research Site 1226, San Antonio, Texas
  - Research Site 1053, San Antonio, Texas
  - Research Site 1063, Salt Lake City, Utah
  - Research Site 1230, Salem, Virginia
- Canada (12):
  - Research Site 5013, Vancouver, British Columbia
  - Research Site 5015, Cambridge, Ontario
  - Research Site 5005, Greater Sudbury, Ontario
  - Research Site 5012, Hamilton, Ontario
  - Research Site 5023, London, Ontario
  - Research Site 5016, Peterborough, Ontario
  - Research Site 5022, Toronto, Ontario
  - Research Site 5014, Toronto, Ontario
  - Research Site 5008, Gatineau, Quebec
  - Research Site 5007, Saint-Charles-Borromée, Quebec
  - Research Site 5009, Saint-Georges, Quebec
  - Research Site 5006, Québec
- Czechia (15):
  - Research Site 3116, Benešov
  - Research Site 3106, Brandýs nad Labem
  - Research Site 3107, Brno
  - Research Site 3118, Brno
  - Research Site 3109, Český Krumlov
  - Research Site 3114, Havířov
  - Research Site 3103, Hradec Králové
  - Research Site 3110, Krnov
  - Research Site 3102, Kroměříž
  - Research Site 3105, Mariánské Lázně
  - Research Site 3113, Pilsen
  - Research Site 3104, Prague
  - Research Site 3111, Prague
  - Research Site 3112, Prague
  - Research Site 3115, Uherské Hradiště
- Denmark (3):
  - Research Site 6104, Copenhagen
  - Research Site 6103, Copenhagen
  - Research Site 6105, Copenhagen
- Mexico (9):
  - Research Site 2015, Guadalajara, Jalisco
  - Research Site 2013, Culiacán, Sinaloa
  - Research Site 2008, Tampico, Tamaulipas
  - Research Site 2012, Mérida, Yucatán
  - Research Site 2011, Aguascalientes
  - Research Site 2009, Chihuahua City
  - Research Site 2014, México
  - Research Site 2016, Querétaro
  - Research Site 2010, Veracruz
- Netherlands (7):
  - Research Site 5101, 's-Hertogenbosch
  - Research Site 5110, Amsterdam
  - Research Site 5113, Harderwijk
  - Research Site 5112, Hoofddorp
  - Research Site 5102, Hoogeveen
  - Research Site 5106, Rotterdam
  - Research Site 5103, Zwijndrecht
- Poland (19):
  - Research Site 7122, Aleksandrów Łódzki
  - Research Site 7113, Gdansk
  - Research Site 7119, Gdynia
  - Research Site 7109, Grodzisk Mazowiecki
  - Research Site 7115, Katowice
  - Research Site 7106, Katowice
  - Research Site 7121, Katowice
  - Research Site 7111, Kutno
  - Research Site 7104, Lodz
  - Research Site 7135, Lodz
  - Research Site 7120, Lublin
  - Research Site 7118, Otwock
  - Research Site 7108, Oława
  - Research Site 7107, Puławy
  - Research Site 7105, Sobótka
  - Research Site 7112, Sochaczew
  - Research Site 7123, Warsaw
  - Research Site 7117, Warsaw
  - Research Site 7116, Warsaw
- Russia (12):
  - Research Site 9309, Lomonosov
  - Research Site 9303, Moscow
  - Research Site 9315, Moscow
  - Research Site 9314, Novosibirsk
  - Research Site 9318, Novosibirsk
  - Research Site 9301, Novosibirsk
  - Research Site 9310, Saint Petersburg
  - Research Site 9304, Saint Petersburg
  - Research Site 9307, Saint Petersburg
  - Research Site 9311, Saint Petersburg
  - Research Site 9312, Saint Petersburg
  - Research Site 9302, Tomsk
- South Korea (7):
  - Research Site 7007, Chuncheon, Gangwon-do
  - Research Site 7001, Wŏnju, Gangwon-do
  - Research Site 7004, Anyang-si, Gyeonggi-do
  - Research Site 7005, Guri-si, Gyeonggi-do
  - Research Site 7006, Busan
  - Research Site 7002, Gwangju
  - Research Site 7008, Incheon
- Taiwan (7):
  - Research Site 8001, Kaohsiung City
  - Research Site 8002, New Taipei City
  - Research Site 8006, Taichung
  - Research Site 8005, Tainan
  - Research Site 8007, Taipei
  - Research Site 8004, Taipei
  - Research Site 8003, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1700 patients were recruited from 10 countries: Canada, Czech Republic, Demark, Republic of Korea, Mexico, the Netherlands, Poland, Russian Federation, Taiwan, and the United States.
Pre-assignment Details: Subjects ≥ 40 years old with inadequately controlled T2DM with HbA1c between 7.5% (7.0% since protocol version 8) and 11% on stable medications and elevated risk for CV adverse events were enrolled. All subjects must belong to 1 of 3 CV risk groups to be eligible. All eligible subjects took placebo during 13 ± 2 days run-in period.
Period: Completed the Study Through Week 24
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Started | 1133 | 567
Completed | 1089 | 542
Not Completed | 44 | 25
Not completed — Adverse Event | 9 | 3
Not completed — Death | 7 | 7
Not completed — Lost to Follow-up | 8 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 17 | 13
Not completed — The subject was randomized, but did not take any investigational product | 1 | 0
Period: Completed the Study
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Started (The number of participants started is equal to ITT population) | 1133 | 567
Completed | 987 | 482
Not Completed | 146 | 85
Not completed — Adverse Event | 14 | 5
Not completed — Death | 39 | 25
Not completed — Lost to Follow-up | 31 | 23
Not completed — Physician Decision | 6 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 53 | 31
Not completed — The subject was randomized, but did not take any investigational product | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets | Total
Number analyzed (Participants) | 1133 | 567 | 1700
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 562 | 276 | 838
  >=65 years | 571 | 291 | 862
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.94) | 64.6 (8.01) | 64.4 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341 | 177 | 518
  Male | 792 | 390 | 1182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 166 | 93 | 259
  Not Hispanic or Latino | 967 | 474 | 1441
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 98 | 54 | 152
  Asian | 108 | 55 | 163
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 46 | 28 | 74
  White | 879 | 430 | 1309
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 67 | 24 | 91
  Netherlands | 36 | 18 | 54
  South Korea | 48 | 26 | 74
  United States | 397 | 205 | 602
  Czechia | 118 | 52 | 170
  Taiwan | 46 | 20 | 66
  Denmark | 17 | 10 | 27
  Poland | 196 | 97 | 293
  Mexico | 121 | 62 | 183
  Russia | 87 | 53 | 140
Cardiovascular Risk Groups [Count of Participants; unit: Participants] — 1: History of atherosclerotic vascular disease with > 1 of the following: i) MI/ischemic stroke > 3 months but < 5 years prior to screening ii) Documented history of coronary, carotid or peripheral arterial revascularization (CABG must have occurred > 5 years prior to screening) 2: History of heart failure 3: Age >= 55 with > 2 of the following: i) Diabetes duration of > 10 years ii) Uncontrolled hypertension defined as SBP > 140 mmHg despite > 3 anti-hypertensive medications iii) current smoker iv) Urine albumin: creatinine ratio > 30 mg/g v) eGFR 45-60 mL/min/1.73 m2 vi) HDL < 1 mmol/L
  Participants
    Group 1: History of atherosclerotic vascular disease | 703 | 362 | 1065
    Group 2: History of heart failure | 166 | 80 | 246
    Group 3: Age >= 55 years with > 2 risk factors | 264 | 125 | 389
Body Weight [Mean (Standard Deviation); unit: kg] | 94.59 (21.87) | 92.62 (19.999) | 93.94 (20.745)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.80 (6.068) | 32.24 (5.751) | 32.62 (5.968)
Body Mass Index Categories [Count of Participants; unit: Participants]
  BMI < 25 kg/m^2 | 86 | 45 | 131
  BMI >= 25 kg/m^2 | 1047 | 522 | 1569
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 134.2 (16.24) | 133.7 (16.18) | 134.0 (16.21)
Systolic Blood Pressure Groups [Count of Participants; unit: Participants]
  < 140 mmHg | 685 | 352 | 1037
  >= 140 mmHg | 448 | 215 | 663
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 77.1 (9.94) | 76.8 (10.16) | 77.0 (10.01)
eGFR at Screening [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 77.93 (19.475) | 77.76 (19.653) | 77.88 (19.529)
eGFR group [Count of Participants; unit: Participants]
  < 60 mL/min/1.73 m^2 | 225 | 109 | 334
  >= 60 mL/min/1.73 m^2 | 908 | 458 | 1366
HbA1c [Mean (Standard Deviation); unit: % of HbA1c] | 8.32 (0.897) | 8.33 (0.944) | 8.32 (0.913)
HbA1c group [Count of Participants; unit: Participants]
  <= 8.5% | 716 | 362 | 1078
  > 8.5% | 417 | 205 | 622
Duration of Diabetes from Diagnosis to the date of informed consent [Mean (Standard Deviation); unit: years] | 14.87 (8.635) | 15.23 (9.253) | 14.99 (8.845)
Insulin Use at Baseline [Count of Participants; unit: Participants]
  Yes | 610 | 292 | 902
  No | 523 | 275 | 798
Use of Anti-Diabetic Treatment at Baseline [Count of Participants; unit: Participants]
  Yes | 1125 | 564 | 1689
  No | 8 | 3 | 11
NT-proBNP [Mean (Standard Deviation); unit: pmol/L] | 391.9 (760.75) | 264.0 (427.15) | 346.1 (661.93)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: % of Left Ventricular Ejection Fraction] | 49.2 (14.13) | 50.8 (12.95) | 49.8 (13.74)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Description: The primary efficacy objective of this trial is to evaluate the placebo-adjusted change in HbA1c from baseline after 24 weeks of treatment with 20 mg bexagliflozin tablets in type 2 diabetic subjects with increased risk of cardiovascular adverse events.
Time Frame: 24 weeks
Population: Number of subjects with a value at baseline and at Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 1046 | 531
percentage of glycated hemoglobin | -0.85 [-0.90 to -0.80] | -0.37 [-0.44 to -0.30]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the primary endpoint was that the mean change in HbA1c from baseline to Week 24 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Superiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 24 was less than the mean change in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; Region, baseline eGFR categories and BMI, history of heart failure, insulin use (Y/N), treatment, visit and baseline HbA1c as fixed effect covariate; Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.56 to -0.39]

2. Secondary Outcome: Change From Baseline in HbA1c at Week 24 for Subjects Who Have Been Prescribed Insulin
Description: To evaluate the effect of 20 mg bexagliflozin on the change in HbA1c from baseline to week 24 in randomized subjects who have been prescribed insulin to control their diabetes
Time Frame: 24 weeks
Population: Number of subjects with a value at baseline and at week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of HbA1c
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 561 | 273
Percentage of HbA1c | -0.84 [-0.92 to -0.77] | -0.32 [-0.43 to -0.22]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the secondary endpoint was that the mean change in HbA1c from baseline to Week 24 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; Region, baseline eGFR categories, history of heart failure, treatment, visit and baseline HbA1c as fixed effect covariate; Mean Difference (Net) = -0.52, 95% CI 2-sided [-0.65 to -0.40]

3. Secondary Outcome: Change in Body Weight From Baseline to Week 48
Description: To evaluate the effect of 20 mg bexagliflozin on the change in body weight from baseline to week 48 in randomized subjects with a BMI ≥ 25 kg/m2 compared to placebo
Time Frame: 48 weeks
Population: Number of subjects with a value at baseline and at Week 48 is included.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 922 | 456
kg | -3.03 [-3.27 to -2.80] | -0.38 [-0.72 to -0.04]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the secondary endpoint was that the mean change in body weight from baseline to Week 48 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Superiority — Rejection of the null hypothesis would imply that the mean change in body weight from baseline to Week 48 was less than the mean change in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; Region, baseline HbA1c and eGFR, history of heart failure, insulin use (Y/N), treatment, visit and baseline body weight as fixed effect covariate; Mean Difference (Net) = -2.65, 95% CI 2-sided [-3.07 to -2.24]

4. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 24 in Subjects Hypertensive at Baseline
Description: To evaluate the effect of 20 mg bexagliflozin on the change in systolic blood pressure (SBP) from baseline to week 24 in subjects with baseline systolic blood pressure ≥ 140 mmHg compared to placebo
Time Frame: 24 weeks
Population: Number of subjects with a value at baseline and at week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 417 | 204
mm Hg | -9.83 [-11.28 to -8.38] | -6.87 [-8.95 to -4.78]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the secondary endpoint was that the mean change in systolic blood pressure from baseline to Week 24 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Superiority — Rejection of the null hypothesis would imply that the mean change in systolic blood pressure from baseline to Week 24 was less than the mean change in the placebo arm by a value that could not be attributed to chance alone; p = 0.0112, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; Region, baseline HbA1c, GFR categories, BMI, history of heart failure, insulin use (Y/N), treatment, visit and baseline SBP as fixed effect covariate; Mean Difference (Net) = -2.96, 95% CI 2-sided [-5.51 to -0.42]

5. Other Pre Specified Outcome: Change in HbA1c From Baseline Over Time
Description: To assess the effect of 20 mg bexagliflozin treatment on the change in HbA1c from baseline versus placebo over time up to 168 weeks
Time Frame: Baseline (week 0) and weeks 6, 12, 24, 36, 48, 72, 96, 120, 144 and 168
Population: Number of subjects with a value at baseline and at the specified visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of HbA1c
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 1133 | 567
Percentage of HbA1c
  Week 6: number analyzed (Participants) | 1111 | 553
  Week 6 | -0.69 [-0.72 to -0.65] | -0.24 [-0.28 to -0.19]
  Week 12: number analyzed (Participants) | 1075 | 544
  Week 12 | -0.89 [-0.94 to -0.85] | -0.34 [-0.39 to -0.28]
  Week 24: number analyzed (Participants) | 1046 | 531
  Week 24 | -0.84 [-0.89 to -0.79] | -0.37 [-0.45 to -0.30]
  Week 36: number analyzed (Participants) | 1017 | 511
  Week 36 | -0.86 [-0.92 to -0.81] | -0.39 [-0.47 to -0.32]
  Week 48: number analyzed (Participants) | 992 | 496
  Week 48 | -0.84 [-0.90 to -0.79] | -0.38 [-0.46 to -0.30]
  Week 72: number analyzed (Participants) | 965 | 469
  Week 72 | -0.76 [-0.83 to -0.70] | -0.34 [-0.44 to -0.25]
  Week 96: number analyzed (Participants) | 874 | 426
  Week 96 | -0.68 [-0.75 to -0.62] | -0.29 [-0.39 to -0.20]
  Week 120: number analyzed (Participants) | 768 | 364
  Week 120 | -0.65 [-0.73 to -0.58] | -0.22 [-0.33 to -0.11]
  Week 144: number analyzed (Participants) | 445 | 196
  Week 144 | -0.62 [-0.71 to -0.53] | -0.23 [-0.37 to -0.10]
  Week 168: number analyzed (Participants) | 218 | 99
  Week 168 | -0.56 [-0.67 to -0.45] | -0.29 [-0.46 to -0.13]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 6 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Superiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 6 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.50 to -0.39]
Statistical Analysis 2: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 12 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 12 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.63 to -0.49]
Statistical Analysis 3: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 24 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 24 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.56 to -0.38]
Statistical Analysis 4: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 36 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 36 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.56 to -0.38]
Statistical Analysis 5: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 48 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 48 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.56 to -0.37]
Statistical Analysis 6: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 72 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 72 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.54 to -0.31]
Statistical Analysis 7: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 96 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 96 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.51 to -0.27]
Statistical Analysis 8: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 120 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 120 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.56 to -0.30]
Statistical Analysis 9: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 144 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 144 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.54 to -0.23]
Statistical Analysis 10: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in HbA1c from baseline to Week 168 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline HbA1c from baseline to Week 168 was less than that in the placebo arm by a value that could not be attributed to chance alone; p = 0.0045, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.47 to -0.07]

6. Other Pre Specified Outcome: Change in Fasting Plasma Glucose Over Time
Description: To evaluate the effect of bexagliflozin treatment on the change in fasting plasma glucose (FPG) versus placebo over time up to 168 weeks
Time Frame: Baseline (week 0) and weeks 6, 12, 24, 36, 48, 72, 96, 120, 144 and 168
Population: Number of subjects with a value at baseline and at the specified visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 1133 | 567
mmol/L
  Week 6: number analyzed (Participants) | 1107 | 552
  Week 6 | -1.28 [-1.40 to -1.16] | 0.07 [-0.10 to 0.24]
  Week 12: number analyzed (Participants) | 1078 | 545
  Week 12 | -1.33 [-1.46 to -1.21] | 0.06 [-0.12 to 0.23]
  Week 24: number analyzed (Participants) | 1045 | 530
  Week 24 | -1.43 [-1.56 to -1.30] | -0.05 [-0.23 to 0.13]
  Week 36: number analyzed (Participants) | 1016 | 513
  Week 36 | -1.21 [-1.36 to -1.06] | -0.06 [-0.27 to 0.15]
  Week 48: number analyzed (Participants) | 996 | 494
  Week 48 | -1.36 [-1.50 to -1.21] | -0.12 [-0.33 to 0.08]
  Week 72: number analyzed (Participants) | 966 | 469
  Week 72 | -1.14 [-1.30 to -0.98] | -0.15 [-0.38 to 0.07]
  Week 96: number analyzed (Participants) | 873 | 425
  Week 96 | -1.16 [-1.32 to -0.99] | 0.04 [-0.20 to 0.29]
  Week 120: number analyzed (Participants) | 765 | 365
  Week 120 | -0.90 [-1.09 to -0.71] | 0.25 [-0.02 to 0.53]
  Week 144: number analyzed (Participants) | 445 | 195
  Week 144 | -1.03 [-1.24 to -0.81] | -0.40 [-0.72 to -0.08]
  Week 168: number analyzed (Participants) | 218 | 101
  Week 168 | -1.06 [-1.39 to -0.73] | -0.55 [-1.04 to -0.07]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 6 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 6 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; Region, baseline eGFR categories & BMI, history of HF, insulin use, treatment, visit, hypoglycemic use and baseline FPG as fixed effect covariate; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-1.55 to -1.15]
Statistical Analysis 2: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 12 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 12 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-1.61 to -1.18]
Statistical Analysis 3: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 24 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 24 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-1.61 to -1.16]
Statistical Analysis 4: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 36 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 36 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.41 to -0.89]
Statistical Analysis 5: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 48 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 48 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.48 to -0.98]
Statistical Analysis 6: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 72 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 72 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-1.27 to -0.72]
Statistical Analysis 7: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 96 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 96 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.50 to -0.90]
Statistical Analysis 8: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 120 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 120 was less than that in the placebo arm by a value that could not be attributed to chance alone; p < 0.0001, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.49 to -0.82]
Statistical Analysis 9: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 144 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 144 was less than that in the placebo arm by a value that could not be attributed to chance alone; p = 0.0008, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.01 to -0.24]
Statistical Analysis 10: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; The null hypothesis for the exploratory endpoint was that the mean change in FPG from baseline to Week 168 in the bexagliflozin arm would be equal to or greater than the mean change in the placebo arm; Test type: Non-Inferiority — Rejection of the null hypothesis would imply that the mean change in baseline FPG from baseline to Week 168 was less than that in the placebo arm by a value that could not be attributed to chance alone; p = 0.0462, Mixed-effects repeated measures — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.09 to 0.08]

7. Other Pre Specified Outcome: Proportion of Subjects Requiring an Intensification of Hypoglycemic Agent and Time to First Intensification
Description: To measure the proportion of subjects requiring an intensification of hypoglycemic agent in the bexagliflozin arm versus placebo during 24 week period
Time Frame: 24 week
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 1133 | 567
Proportion of participants | 0.06 [0.05 to 0.08] | 0.18 [0.15 to 0.21]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value is based on one sided statistical tests using a 0.025 level of significance; Region, baseline eGFR categories & BMI, history of heart failure, insulin use (Y/N), treatment and baseline HbA1c as fixed effect covariate; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.22 to 0.41] — Odds ratio is calculated as the odds ratio of bexagliflozin over placebo

8. Other Pre Specified Outcome: Proportion of Subjects Requiring an Intensification of Hypoglycemic Agent and Time to First Intensification
Description: To measure the proportion of subjects requiring an intensification of hypoglycemic agent in the bexagliflozin arm versus placebo during the entire study period
Time Frame: Duration of study (168 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 1133 | 567
Proportion of participants | 0.06 [0.05 to 0.08] | 0.18 [0.15 to 0.21]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p < 0.0001, Regression, Cox — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.35 to 0.49] — Hazard ratio and p-value were estimated using Cox regression model for time to first event in the bexagliflozin arm vs. placebo arm during entire study

9. Other Pre Specified Outcome: Proportion of Subjects Requiring a Relaxation of Hypoglycemic Agent
Description: To measure the proportion of subjects requiring a relaxation of hypoglycemic agent in the bexagliflozin arm versus placebo during 24 week period
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 1133 | 567
Proportion of participants | 0.09 [0.08 to 0.11] | 0.05 [0.03 to 0.07]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p = 0.0005, Regression, Logistic — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.33 to 3.11] — Odds ratio is calculated as the ratio of bexagliflozin over placebo

10. Other Pre Specified Outcome: Proportion of Subjects Requiring a Relaxation of Hypoglycemic Agent
Description: To measure the proportion of subjects requiring a relaxation of hypoglycemic agent in the bexagliflozin arm versus placebo during the entire study
Time Frame: Duration of study (168 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
Number analyzed (Participants) | 1133 | 567
Proportion of participants | 0.09 [0.08 to 0.11] | 0.05 [0.03 to 0.07]
Statistical Analysis 1: Comparison: Bexagliflozin Tablets, 20 mg vs Placebo Tablets; Test type: Superiority; p < 0.0001, Regression, Cox — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.82, 95% CI 2-sided [1.40 to 2.38] — Hazard ratio and p-value were estimated using Cox regression model for time to first event in the bexagliflozin arm vs. placebo arm during the entire study

11. Other Pre Specified Outcome: Proportion of Participants With Incidence of Hospitalization for Heart Failure
Description: To measure the incidence of hospitalization for heart failure among all subjects and among subjects who have a history of heart failure at baseline
Time Frame: Duration of study (168 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- All Subjects: Bexagliflozin Tablets, 20 mg: Each subject will receive bexagliflozin 20 mg once daily for the duration of the study.
  Bexagliflozin: 20 mg, tablet
  This group includes all subjects who have received bexagliflozin in the study.
- All Subjects: Placebo Tablets: Each subject will receive placebo (inactive tablet) once daily for the duration of the study.
  Placebo: 20 mg tablet to match active comparator
  This group includes all subjects who have received placebo in the study.
- Subjects With HF History: Bexagliflozin Tablets, 20 mg: Each subject will receive bexagliflozin 20 mg once daily for the duration of the study.
  Bexagliflozin: 20 mg, tablet
  This group includes subjects who reported a history of heart failure and randomized to the bexagliflozin arm.
- Subjects With HF History: Placebo: Each subject will receive placebo (inactive tablet) once daily for the duration of the study.
  Placebo: 20 mg tablet to match active comparator
  This group includes subjects who reported a history of heart failure and randomized to the placebo arm.
Arm/Group | All Subjects: Bexagliflozin Tablets, 20 mg | All Subjects: Placebo Tablets | Subjects With HF History: Bexagliflozin Tablets, 20 mg | Subjects With HF History: Placebo
Number analyzed (Participants) | 1133 | 567 | 302 | 151
Proportion of participants | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.03] | 0.05 [0.03 to 0.08] | 0.09 [0.05 to 0.15]
Statistical Analysis 1: Comparison: All Subjects: Bexagliflozin Tablets, 20 mg vs All Subjects: Placebo Tablets; Test type: Superiority; p = 0.0803, Regression, Logistic — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.33 to 1.20] — Odds ratio is calculated as the odds ratio of bexagliflozin over placebo
Statistical Analysis 2: Comparison: Subjects With HF History: Bexagliflozin Tablets, 20 mg vs Subjects With HF History: Placebo; Test type: Superiority; p = 0.0272, Regression, Logistic — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.22 to 1.01] — Odds ratio is calculated as the odds ratio of bexagliflozin over placebo
Statistical Analysis 3: Comparison: All Subjects: Bexagliflozin Tablets, 20 mg vs All Subjects: Placebo Tablets; Test type: Superiority; p = 0.0757, Regression, Cox — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.34 to 1.18] — Hazard ratio and p-value were estimated using Cox regression model for treatment comparison vs. placebo
Statistical Analysis 4: Comparison: Subjects With HF History: Bexagliflozin Tablets, 20 mg vs Subjects With HF History: Placebo; Test type: Superiority; p = 0.0273, Regression, Cox — P-value is based on one sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.23 to 1.01] — Hazard ratio and p-value were estimated using Cox regression model for treatment comparison vs. placebo

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first dose to the last day of follow up (4 weeks after the End of Treatment visit, an average of 127 weeks)
Arm/Group | Bexagliflozin Tablets, 20 mg | Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 39/1132 | 26/567
Serious Adverse Events (participants affected / at risk) | 373/1132 | 208/567
Other Adverse Events (participants affected / at risk) | 739/1132 | 386/567
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin Tablets, 20 mg (N=1132) | Placebo Tablets (N=567)
Angina unstable (Cardiac disorders) | 31 (39) | 19 (22)
Acute myocardial infarction (Cardiac disorders) | 31 (33) | 14 (15)
Cardiac failure congestive (Cardiac disorders) | 18 (21) | 15 (21)
Cardiac failure (Cardiac disorders) | 21 (27) | 7 (9)
Angina pectoris (Cardiac disorders) | 16 (20) | 11 (12)
Coronary artery disease (Cardiac disorders) | 21 (21) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 15 (21) | 9 (17)
Myocardial infarction (Cardiac disorders) | 11 (11) | 13 (13)
Cardiac arrest (Cardiac disorders) | 12 (12) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 5 (6) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 8 (8) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 6 (7)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 3 (3)
Atrial flutter (Cardiac disorders) | 3 (3) | 2 (4)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Anginal equivalent (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (3) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 11 (11) | 10 (10)
Cellulitis (Infections and infestations) | 9 (11) | 2 (2)
Osteomyelitis (Infections and infestations) | 10 (13) | 1 (1)
Sepsis (Infections and infestations) | 9 (9) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (3)
Gangrene (Infections and infestations) | 4 (5) | 3 (4)
Diverticulitis (Infections and infestations) | 3 (3) | 3 (3)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Localised infection (Infections and infestations) | 4 (4) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 1 (1)
Endocarditis (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Medical device site joint infection (Infections and infestations) | 1 (1) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 15 (15) | 7 (7)
Ischaemic stroke (Nervous system disorders) | 10 (11) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 6 (7) | 5 (6)
Carotid artery stenosis (Nervous system disorders) | 7 (9) | 3 (3)
Syncope (Nervous system disorders) | 4 (4) | 4 (4)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Miller Fisher syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 11 (12) | 7 (8)
Peripheral arterial occlusive disease (Vascular disorders) | 8 (11) | 6 (8)
Hypotension (Vascular disorders) | 5 (5) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 3 (3) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2)
Intermittent claudication (Vascular disorders) | 1 (3) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 2 (3) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (2)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 (17) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Immunoglobulin G4 related sclerosing disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barret's oesophagus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 3 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 3 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 14 (15) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 6 (7) | 5 (5)
Chest pain (General disorders) | 6 (7) | 3 (3)
Necrosis (General disorders) | 3 (3) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 9 (10) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 3 (4) | 2 (2)
Calculus ureteric (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cervix disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (4) | 1 (1)
Corneal lesion (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Keratopathy (Eye disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin Tablets, 20 mg (N=1132) | Placebo Tablets (N=567)
Diarrhoea (Gastrointestinal disorders) | 72 (90) | 31 (40)
Nausea (Gastrointestinal disorders) | 54 (64) | 37 (45)
Bronchitis (Infections and infestations) | 52 (65) | 34 (40)
Nasopharyngitis (Infections and infestations) | 96 (115) | 39 (46)
Upper respiratory tract infection (Infections and infestations) | 112 (147) | 53 (82)
Urinary tract infection (Infections and infestations) | 128 (190) | 60 (96)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 49 (53) | 29 (37)
Hyperglycaemia (Metabolism and nutrition disorders) | 68 (181) | 41 (80)
Hypoglycaemia (Metabolism and nutrition disorders) | 475 (3743) | 246 (1857)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (56) | 30 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 66 (72) | 33 (36)
Hypertension (Vascular disorders) | 45 (46) | 36 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT02558296/Prot_SAP_000.pdf